CLINICAL TRIAL: NCT05044520
Title: Clinical Features Associated With Restless Legs Syndrome : Clin-RLS
Brief Title: Clinical Features Associated With Restless Legs Syndrome.
Acronym: Clin-RLS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0535
Record Dates: First submitted 2021-09-06; First posted 2021-09-14 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Restless Legs Syndrome
Keywords: Restless legs syndrome; Augmentation syndrome; Dopamine agonists; Alpha 2 delta ligands; Opiates
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Restless legs syndrome (RLS) is a chronic neurological disorder characterized by an urge to move the legs at night when at rest. RLS can lead to a sleep deprivation, increased falling risk, daytime sleepiness, depression and decreased quality of life. Dopamine agonists, alpha-2-delta ligands and opiates are key medications for RLS. The natural course of RLS is very heterogeneous with a risk of increasing the severity of symptoms over the years despite the use of drugs and recommended dosages. Many comorbidities can make RLS worse. Augmentation syndrome is the main complication of dopamine agonists. However, only a few studies have addressed the clinical, biological and pharmacological factors associated with the evolution of the severity of RLS. The objective of this study is to assess the evolution of RLS symptoms severity as function of RLS phenotype, comorbidities and RLS medication, in large cohort of members of the French RLS association and other European RLS association.

DETAILED DESCRIPTION:
In this study, the investigators want to study the clinical course of RLS in a population of RLS patients who are members of the RLS patient association, taking into account clinical and biological factors as well as the treatments taken for RLS.

ELIGIBILITY:
Inclusion criteria:

* Adults subjects
* Restless legs syndrome diagnosis
* Member of the restless legs syndrome association
* French speaking
* Able to understand the study
* Signed written informed consent
* Affiliated to social security

Exclusion criteria:

- Vulnerable subject : subject deprived of liberty or protected by law (trusteeship, legal guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RLS who are members of the RLS patient association
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
International restless legs syndrome study group rating scale (IRLS) | Four minutes
  International restless legs syndrome study group rating scale (IRLS). ranging from 0 to 40, with higher scores indicating worse restless legs symptoms

SECONDARY OUTCOMES:
Restless Legs Syndrome-6 Scale (RLS-6) | two minutes
  Restless Legs Syndrome-6 Scale (RLS-6)symptoms after a surgical procedure under general or locoregional anesthesia. ranging from 0 to 60, with higher scores indicating worse restless legs symptoms
Augmentation Severity Rating Scale (ASRS) | two minutes
  Augmentation Severity Rating Scale (ASRS). ranging from 0 to 24, with higher scores indicating worse augmentation symptoms
Epworth severity scale (ESS) | two minutes
  Epworth severity scale (ESS). ranging from 0 to 24, with higher scores indicating worse sleepiness
Insomnia Severity Index (ISI) | two minutes
  Insomnia Severity Index (ISI). ranging from 0 to 28, with higher scores indicating worse insomnia
Beck's Depression Inventory - II (BDI-II) | Six minute
  Beck's Depression Inventory - II (BDI-II). ranging from 0 to 63, with higher scores indicating worse depressive symptoms
European Quality of life - 5 dimensions (EQ-5D) | One minute
  European Quality of life - 5 dimensions (EQ-5D). ranging from 0 to 100. Higher scores indicate better health condition
Homemade questionnaire assessing the falling risk | Five minutes
  Homemade questionnaire assessing the falling risk. ranging from 0 to 6, with higher scores indicating worse falling risk

CONTACTS AND LOCATIONS:
Overall Officials: Yves DAUVILLIERS, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC